CLINICAL TRIAL: NCT02580149
Title: The Effect of an Acute Dose of Ticagrelor or Clopidogrel and of Treatment for 14 Days on Ischemia-reperfusion Induced Endothelial Dysfunction of the Forearm Vasculature in Healthy Male Subjects.
Brief Title: The Effect of Ticagrelor or Clopidogrel on Endothelial Function During Acute and Chronic Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michael Wolzt, Prof. MD (Other)
Responsible Party: Sponsor-Investigator, Michael Wolzt, Prof. MD, Prof. MD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FBF-Tica-Clopi
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Ischemia
MeSH Terms: conditions — Ischemia | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Active Comparator): Loading dose of 180 mg on day one, followed by a regular intake (90 mg twice daily) for 14 days
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): Loading dose of 600 mg on day one, followed by a regular intake (75 mg once daily) for 14 days
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Subjects will receive an oral loading dose of 180 mg ticagrelor on study day
  1 followed by a maintenance dose of 90 mg twice daily for 14 days (until study day 15).
  Other Names: Brilique
  Arms: Ticagrelor
Drug: Clopidogrel — Subjects will receive a loading dose of 600 mg clopidogrel on the first study day followed by a maintenance dose of 75 mg once daily for 14 days
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
To investigate if treatment with ticagrelor can mitigate the transient loss of endothelium-dependent vasodilatation of the resistance vasculature following a short period of ischemia, compared with clopidogrel at standard clinical doses. The effect of ticagrelor or clopidogrel will be studied after a loading dose and after a two weeks period of regular intake on FBF in response to the vasodilators acetylcholine or nitroglycerin before and 10 min after a 20 min forearm ischemia, respectively.

DETAILED DESCRIPTION:
Ischemia-reperfusion (IR) causes tissue injury. Preclinical animal data suggest that ticagrelor but not clopidogrel protects against IR injury due to inhibition of cellular adenosine uptake and NO-synthase stimulation. It is unclear if this action is part of the beneficial clinical effect of ticagrelor in patients with a history of acute coronary syndrome. The preventive action of ticagrelor on IR injury may also be of interest for the peripheral vasculature, where IR injury is known to result in endothelial dysfunction. This study aims to investigate if treatment with ticagrelor can mitigate the transient loss of endothelium-dependent vasodilatation of the resistance vasculature following a short period of ischemia, compared with clopidogrel at standard clinical doses. We will study the effect of ticagrelor or clopidogrel after a loading dose and after a two weeks period of regular intake on forearm blood flow (FBF) reactivity in response to the vasodilators acetylcholine (ACh; endothelium-dependent agonist) or nitroglycerin (GTN; endothelium-independent vasodilator) before and 10 min after a 20 min forearm ischemia, respectively

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects; 18 - 40 years of age
* Body mass index between 18 and 27 kg/m2
* Written informed consent
* Normal findings in medical & bleeding history
* Non-smoking

Exclusion Criteria:

* Regular intake of any medication including OTC drugs and herbals within 2 weeks before IMP administration
* Known coagulation disorders (e.g. haemophilia, von Willebrand´s disease)
* Known disorders with increased bleeding risk (e.g. peridontosis, haemorrhoids, acute gastritis, peptic ulcer, intestinal ulcer)
* Known sensitivity to common causes of bleeding (e.g. nasal)
* History of thromboembolism
* History of occlusive vascular diseases
* History of vascular anomalies
* Impaired liver function (AST, ALT, gGT, bilirubin >2 x ULN)
* Impaired renal function (serum creatinine > 1.3 mg/dl)
* Any other relevant deviation from the normal range in clinical chemistry, haematology or urine analysis
* HIV-1/2-Ab, HbsAg or HCV-Ab positive serology
* Systolic blood pressure above 145 mmHg, diastolic blood pressure above 95 mmHg
* Known allergy against any test agent under study
* Regular daily consumption of more than on litre of xanthine-containing beverages or more than 40g alcohol
* Participation in another clinical trial during the preceding 3 weeks

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of Forearm blood flow (FBF) measurements of Acetylcholin (ACh) induced vasodilatation | Change of the AUC before and 10 min after forearm ischemia
  To test the effect of ticagrelor or clopidogrel on ACh-induced vasodilatation of the forearm resistance vasculature as assessed by FBF measurement before and 10 min after a 20 min forearm ischemia.

SECONDARY OUTCOMES:
Area under the curve (AUC) of Forearm blood flow (FBF) measurements of Glyceroltrinitrate (GTN) induced vasodilatation | Change of AUC before and 10 min after forearm ischemia
  To test the effect of ticagrelor or clopidogrel on GTN-induced vasodilatation of the forearm resistance vasculature as assessed by FBF measurement before and 10 min after a 20 min forearm ischemia.
(Expected) Peak plasma concentration of ticagrelor or clopidogrel | 2.5 h after IMP intake

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, Prof. MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Vienna, Austria